CLINICAL TRIAL: NCT04193176
Title: A Phase 3b Randomized, Double-blind, Placebo Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Gefapixant in Women With Chronic Cough and Stress Urinary Incontinence
Brief Title: Efficacy and Safety of Gefapixant (MK-7264) in Women With Chronic Cough and Stress Urinary Incontinence (MK-7264-042)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7264-042; MK-7264-042 (Other: MSD Protocol Number); 2019-002321-29 (EudraCT Number)
Record Dates: First submitted 2019-12-09; First posted 2019-12-10 (Actual); Results first posted 2023-09-22 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Chronic Cough
Keywords: Cough; Urinary Incontinence, Stress; Respiration disorders; Respiratory tract diseases; Signs and symptoms, respiratory; Signs and symptoms
MeSH Terms: conditions — Chronic Cough; Cough; Urinary Incontinence, Stress; Respiration Disorders; Respiratory Tract Diseases; Signs and Symptoms, Respiratory; Signs and Symptoms | interventions — Gefapixant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gefapixant (Experimental): Participants will receive gefapixant at a dose of 45 mg administered as an oral tablet twice daily for 12 weeks.
  Interventions: Drug: Gefapixant
- Placebo (Placebo Comparator): Participants will receive placebo matching gefapixant, administered as an oral tablet twice daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gefapixant — Administered twice daily as an oral tablet of 45 mg
  Other Names: MK-7264
  Arms: Gefapixant
Drug: Placebo — Administered twice daily as a placebo oral tablet matching gefapixant
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of gefapixant, in improving symptoms of cough-induced stress urinary incontinence (SUI) in adult female participants with refractory or unexplained chronic cough. The primary hypothesis is that gefapixant is superior to placebo in reducing the frequency of cough-induced SUI episodes over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Has a chest radiograph or computed tomography scan of the thorax (within 5 years of Screening and after the onset of chronic cough) not demonstrating any abnormality considered to be significantly contributing to the chronic cough or any other lung disease
* Has chronic cough (defined as duration of >8 weeks after onset of cough symptoms) for ≥12 months
* Has a diagnosis of refractory chronic cough or unexplained chronic cough
* Has symptoms of SUI, defined as involuntary loss of urine on effort, physical exertion, or on sneezing or coughing, for ≥3 months
* Is a female who is not pregnant, not breastfeeding, not of childbearing potential, or agrees to follow contraceptive guidance

Exclusion Criteria:

* Is a current smoker
* Has given up smoking within 12 months of screening
* Is a former smoker with a smoking history greater than 20 pack-years (1 pack of 20 cigarettes per day for 20 years)
* Has a history of respiratory tract infection or recent change in pulmonary status within 4 weeks of screening
* Has a history of chronic bronchitis
* Has a history of surgery to treat SUI within 1 year of screening
* Has a history of other specialized treatments for SUI, including intravesical balloon or urethral bulking agent therapy
* Has other external incontinence device currently or within 1 month of screening
* Has a history of Grade 3 or higher pelvic organ prolapse previously documented or diagnosed on screening
* Has a neurogenic bladder
* Has a history of adult nocturnal incontinence
* Has a history of continuous urine leakage within 1 month of screening
* Has a history of interstitial cystitis
* Has a history of neurological disease or injury
* Has active or recurrent urinary tract infection
* Has a history of having a permanent urinary catheter or any urinary catheterization within 3 months of screening
* Has a history of malignancy ≤5 years prior to signing informed consent
* Is a user of recreational or illicit drugs or a recent history (within the last year) of drug or alcohol abuse
* Has a known allergy to gefapixant or its excipients
* Has donated or lost ≥1 unit (~300 mL) of blood within 8 weeks prior to first dose of gefapixant
* Requires certain medications and/or other therapies that may impact their cough or bladder function
* Has previously received gefapixant
* Is currently participating or has participated in an interventional clinical study within 30 days of participating in this current study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (90):
- United States (19):
  - Center for Clinical Trials, LLC ( Site 0021), Paramount, California
  - Health Awareness, Inc. ( Site 0038), Jupiter, Florida
  - Well Pharma Medical Research, Corp. ( Site 0040), Miami, Florida
  - Lenus Research & Medical Group Llc ( Site 0007), Sweetwater, Florida
  - Florida Pulmonary Research Institute, LLC ( Site 0008), Winter Park, Florida
  - Paul A. Shapero, MD ( Site 0037), Bangor, Maine
  - Chesapeake Clinical Research, Inc ( Site 0022), White Marsh, Maryland
  - University of Missouri ENT & Allergy Center ( Site 0010), Columbia, Missouri
  - Alliance for Multispecialty Research, LLC ( Site 0035), Las Vegas, Nevada
  - Albuquerque Clinical Trials ( Site 0019), Albuquerque, New Mexico
  - American Health Research ( Site 0027), Charlotte, North Carolina
  - Clinical Research of Gastonia ( Site 0016), Gastonia, North Carolina
  - PMG Research of Wilmington ( Site 0004), Wilmington, North Carolina
  - Temple University ( Site 0003), Philadelphia, Pennsylvania
  - AAPRI Clinical Research Institute ( Site 0031), Warwick, Rhode Island
  - Diagnostics Research Group ( Site 0013), San Antonio, Texas
  - TPMG Clinical Research ( Site 0025), Newport News, Virginia
  - Tidewater Physician Multispecialty Group, PC ( Site 0028), Williamsburg, Virginia
  - Bellingham Asthma & Allergy ( Site 0006), Bellingham, Washington
- Argentina (2):
  - Centro Medico Dra De Salvo ( Site 0300), Buenos Aires
  - Investigaciones en Patologias Respiratorias ( Site 0302), San Miguel de Tucumán
- Colombia (4):
  - Fundacion Centro de Investigacion Clinica CIC ( Site 0401), Medellín, Antioquia
  - Universidad Pontificia Bolivariana - Clinica Universitaria Bolivariana ( Site 0408), Medellín, Antioquia
  - Medplus Medicina Prepagada ( Site 0402), Bogotá, Bogota D.C.
  - Healthy Medical Center S.A.S ( Site 0404), Zipaquirá, Cundinamarca
- Germany (5):
  - Praxis Dr. Wehgartner-Winkler ( Site 0906), Augsburg, Bavaria
  - Zentrum fuer ambulante pneumologische Forschung Marburg GbR ( Site 0900), Marburg, Hesse
  - Ballenberger Freytag Wenisch Institut fuer klinische Forschung GmbH ( Site 0905), Neu-Isenburg, Hesse
  - Pneumologicum im Suedstadtforum ( Site 0908), Hanover, Lower Saxony
  - Praxis an der Oper ( Site 0912), Berlin
- Guatemala (6):
  - Bethel Soluciones Medicas S.A. ( Site 0506), Guatemala City
  - Centro de Investigaciones Clinicas de Latinoamerica S.A. - CELAN ( Site 0500), Guatemala City
  - Clinica Medica Especializada en Neumologia y Tisiologia ( Site 0504), Guatemala City
  - Clinica Medica Especializada en Neumologia ( Site 0502), Guatemala City
  - Private Clinic ( Site 0505), Guatemala City
  - Clinica Privada Dr. Jose Francisco Flores Lopez ( Site 0503), Guatemala City
- Israel (7):
  - Carmel Medical Center ( Site 1104), Haifa
  - Shaare Zedek Medical Center ( Site 1107), Jerusalem
  - Hadassah Ein Karem Jerusalem ( Site 1108), Jerusalem
  - Rabin Medical Center ( Site 1102), Petah Tikva
  - Chaim Sheba Medical Center ( Site 1101), Ramat Gan
  - Kaplan Medical Center ( Site 1103), Rehovot
  - Sourasky Medical Center ( Site 1100), Tel Aviv
- Peru (4):
  - Clinica Ricardo Palma ( Site 0601), San Isidro, Lima region
  - Asociacion Civil por la Salud ( Site 0602), Lima
  - Hospital Nacional Arzobispo Loayza ( Site 0607), Lima
  - Clinica Belen ( Site 0604), Piura
- Russia (16):
  - RSBHI Belgorod regional clinical hospital of Prelate Ioasafa ( Site 1416), Belgorod, Belgorod Oblast
  - GBUZ Regional Clinical Hospital 3 ( Site 1420), Chelyabinsk, Chelyabinsk Oblast
  - City Clinical Hospital No. 3 them. M. A. Podgorbunskogo ( Site 1400), Kemerovo, Kemerovo Oblast
  - Open Joint Stock Company Clinical and Diagnostic Center Euromedservice ( Site 1466), Moscow, Moscow
  - Krasnogorsk City Hospital Number 1 ( Site 1470), Krasnogorsk, Moscow Oblast
  - City Clinical Hospital of Emergency Care #2 ( Site 1448), Novosibirsk, Novosibirsk Oblast
  - Clinic of FSBEI HE OmSMU of Minzdrav ( Site 1438), Omsk, Omsk Oblast
  - Perm Clinical Center of the Federal Medical and Biological Agency ( Site 1450), Perm, Permskiy Kray
  - Medi Kom ( Site 1456), Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company Kurator ( Site 1424), Saint Petersburg, Sankt-Peterburg
  - SEIHPE Saint Petersburg SMU ( Site 1434), Saint Petersburg, Sankt-Peterburg
  - Saratov City Clinical Hospital 2 n.a. V.I. Razumovsky ( Site 1452), Saratov, Saratov Oblast
  - Family Clinic ( Site 1464), Yekaterinburg, Sverdlovsk Oblast
  - State health Agency Ulyanovsk regional clinical hospital ( Site 1414), Ulyanovsk, Ulyanovsk Oblast
  - Voronezh Regional Clinical Hospital #1 ( Site 1440), Voronezh, Voronezskaja Oblast
  - SBCIH of the Yaroslavl region Central city hospital ( Site 1428), Yaroslavl, Yaroslavl Oblast
- South Korea (5):
  - Jeonbuk National University Hospital ( Site 1507), Jeonju, Jeonrabugdo
  - Wonju Severance Christian Hospital ( Site 1502), Wŏnju, Kang-won-do
  - The Catholic University of Korea Eunpyeong St Mary s Hospital ( Site 1506), Seoul
  - Konkuk University Medical Center ( Site 1504), Seoul
  - Asan Medical Center ( Site 1505), Seoul
- Spain (4):
  - Hospital Parc Tauli ( Site 1806), Sabadell, Barcelona
  - Hospital Clinic i Provincial de Barcelona ( Site 1804), Barcelona, Catalonia
  - Hospital Clinico Universitario de Santiago ( Site 1805), Santiago de Compostela, La Coruna
  - Hospital General Universitario Gregorio Maranon ( Site 1808), Madrid, Madrid, Comunidad de
- Ukraine (10):
  - F.G.Yanovskyy Institute of Phthisiology and Pulmonology ( Site 2808), Kyiv, Kyivska Oblast
  - F.G.Yanovskyy Institute of Phthisiology and Pulmonology ( Site 2819), Kyiv, Kyivska Oblast
  - SE Road Clinical Hospital 2 of Kyiv station ( Site 2812), Kyiv, Kyivska Oblast
  - SE O.S.Kolomiychenko Institute of Otolaryngology of NAMS of Ukraine ( Site 2817), Kyiv, Kyivska Oblast
  - Odesa regional clinical hospital ( Site 2804), Odesa, Odesa Oblast
  - City Polyclinic N20 ( Site 2806), Odesa, Odesa Oblast
  - Municipal enterprise "1st City clinical hospital of Poltava -Internal medicine department ( Site 281, Poltava, Poltava Oblast
  - Private Small-Scale Enterprise Medical Centre "Pulse" ( Site 2809), Vinnytsia, Vinnytsia Oblast
  - Volyn Regional Clinical Hospital ( Site 2816), Lutsk, Volyn Oblast
  - Medical Center of LLC Medical Clinic Blahomed ( Site 2815), Kyiv
- United Kingdom (8):
  - GP Direct ( Site 2714), Harrow, England
  - West Walk Surgery ( Site 2700), Yate, Gloucestershire
  - Medinova Lakeside Dedicated Research Centre ( Site 2712), Corby, Northamptonshire
  - Kings College Hospital NHS Foundation Trust ( Site 2702), London, Southwark
  - Accellacare South London Quality Research Centre ( Site 2706), Orpington, Surrey
  - Wokingham Medical Centre ( Site 2708), Wokingham, West Berkshire
  - Medinova North London Dedicated Research Centre ( Site 2705), Northwood, Worcestershire
  - Medinova Warwickshire Dedicated Research Centre ( Site 2715), Coventry

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Birring SS, Cardozo L, Dmochowski R, Dicpinigaitis P, Afzal A, La Rosa C, Lu S, Nguyen AM, Yao R, Reyfman PA. Efficacy and safety of gefapixant in women with chronic cough and cough-induced stress urinary incontinence: a phase 3b, randomised, multicentre, double-blind, placebo-controlled trial. Lancet Respir Med. 2024 Nov;12(11):855-864. doi: 10.1016/S2213-2600(24)00222-4. Epub 2024 Aug 30. PMID 39222649
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 376 randomized participants, 375 participants received treatment.
Groups:
- Placebo: Participants received placebo administered as an oral tablet twice daily for 12 weeks.
- Gefapixant: Participants received gefapixant at a dose of 45 mg administered as an oral tablet twice daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Gefapixant
Started | 190 | 186
Treated | 190 | 185
Completed | 184 | 176
Not Completed | 6 | 10
Not completed — Withdrawal by Subject | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Gefapixant | Total
Number analyzed (Participants) | 190 | 186 | 376
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (11.3) | 56.2 (11.5) | 56.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 186 | 376
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 79 | 73 | 152
  Not Hispanic or Latino | 111 | 113 | 224
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 16 | 34
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 143 | 137 | 280
  More than one race | 26 | 24 | 50
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilograms] — Mean weight of participants
  kilograms | 75.6 (13.1) | 75.9 (13.3) | 75.8 (13.2)
Height [Mean (Standard Deviation); unit: centimeters] — Mean height of participants
  centimeters | 159.6 (6.9) | 159.8 (7.0) | 159.7 (7.0)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Mean body mass index of participants
  kg/m^2 | 29.7 (4.4) | 29.7 (4.8) | 29.7 (4.6)
Region [Count of Participants; unit: Participants] — Region of participants
  Participants
    North America | 11 | 9 | 20
    Europe | 102 | 102 | 204
    Asia Pacific | 3 | 3 | 6
    Other | 74 | 72 | 146
Primary cough diagnosis [Count of Participants; unit: Participants] — Primary type of cough diagnosis was categorized as either refractory chronic cough or unexplained chronic cough.
  Participants
    Refractory Chronic Cough | 149 | 141 | 290
    Unexplained Chronic Cough | 41 | 45 | 86
Duration of Chronic Cough [Mean (Standard Deviation); unit: Years] — Duration of chronic cough in years for participants with data Population: Participants with data
  Years
    number analyzed (Participants) | 143 | 155 | 298
    (all) | 5.1 (6.6) | 5.3 (6.5) | 5.2 (6.6)
Baseline Mean Weekly Cough Severity in Visual Analog Scale (VAS) in mm [Mean (Standard Deviation); unit: VAS (mm)] — The Cough Severity VAS is a single-item question asking the participant to rate the severity of their cough "today" using a 100 mm VAS anchored with "No Cough" at 0 and "Extremely Severe Cough" at 100. Similar to the well-established use of VAS scores in chronic pain, the Cough Severity VAS measure provides a quick and easily-interpreted subjective assessment useful for clinicians to monitor improvement of their chronic cough patients following treatment. Baseline mean weekly cough severity in participants measured in Visual Analog Scale in mm is presented. Population: Participants with data
  VAS (mm)
    number analyzed (Participants) | 190 | 185 | 375
    (all) | 69.5 (15.6) | 69.3 (15.8) | 69.4 (15.7)
Duration of Stress Urinary Incontinence (SUI) [Mean (Standard Deviation); unit: Months] — Duration of stress urinary incontinence in participants
  Months | 53.8 (80.8) | 43.4 (58.3) | 48.7 (70.7)
Baseline Mean Daily Cough-Induced Stress Urinary Incontinence Episodes, 7-day Average [Mean (Standard Deviation); unit: Number of episodes] — Baseline Mean Daily Cough-Induced Stress Urinary Incontinence Episodes, 7-day Average for participants Population: Participants who had data
  Number of episodes
    number analyzed (Participants) | 189 | 185 | 374
    (all) | 4.7 (4.1) | 4.7 (3.0) | 4.7 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Average Daily Cough-induced Stress Urinary Incontinence (SUI) Episodes at Week 12
Description: Cough-induced SUI episodes were assessed using an event-driven electronic Incontinence Diary where the participant recorded the main cause of each urinary incontinence episode as coughing, another stress reason, or other cause. Episodes of incontinence were recorded for the week before baseline and treatment visit. Average daily cough induced SUI episodes were calculated as (sum of daily cough-induced SUI episodes in a week)/number of days recorded. The percent change from baseline in the average daily cough-induced SUI episodes to Week 12 are presented.
Time Frame: Baseline and week 12
Population: All randomized participants who received at least 1 dose of study intervention and had incontinence frequency of at least 4 days in the 7-day period prior to the visit at Week 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Gefapixant
Number analyzed (Participants) | 185 | 183
Percent Change | -41.09 [-46.74 to -35.45] | -52.78 [-58.44 to -47.09]
Statistical Analysis 1: Comparison: Placebo vs Gefapixant; Test type: Superiority; p = 0.004, ANCOVA; Mean Difference (Net) = -11.67, 95% CI 2-sided [-19.67 to -3.67]

2. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experienced an adverse event are presented.
Time Frame: Up to ~16 weeks
Population: All randomized participants who received at least one dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Gefapixant
Number analyzed (Participants) | 190 | 185
Percentage of participants | 37.4 | 69.7

3. Secondary Outcome: Percentage of Participants Who Discontinued Study Intervention Due to AEs
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinued study intervention due to an adverse event are presented.
Time Frame: Up to ~14 weeks
Population: All randomized participants who received at least one dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Gefapixant
Number analyzed (Participants) | 190 | 185
Percentage of participants | 1.1 | 7.0

ADVERSE EVENTS:
Time Frame: All deaths and adverse events: up to 16 Weeks
Description: Every participant is counted a single time for each applicable serious adverse event. A system organ class appears on this report only if one or more specific serious adverse events in that system organ class occurred.
Arm/Group | Placebo | Gefapixant
All-Cause Mortality (participants affected / at risk) | 0/190 | 0/186
Serious Adverse Events (participants affected / at risk) | 2/190 | 3/185
Other Adverse Events (participants affected / at risk) | 12/190 | 104/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=190) | Gefapixant (N=185)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=190) | Gefapixant (N=185)
Nausea (Gastrointestinal disorders) | 2 (2) | 10 (10)
Ageusia (Nervous system disorders) | 1 (1) | 35 (36)
Dysgeusia (Nervous system disorders) | 4 (4) | 57 (59)
Headache (Nervous system disorders) | 5 (5) | 13 (14)
Hypogeusia (Nervous system disorders) | 0 (0) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT04193176/Prot_SAP_000.pdf